CLINICAL TRIAL: NCT02807532
Title: Relationship Between Apelin and New-onset Atrial Fibrillation After Coronary Artery Bypass Grafting: a Prospective Cohort Study and Retrospective Case-Control Clinical Trial
Brief Title: Relationship Between Apelin and New-onset Atrial Fibrillation After Coronary Artery Bypass Grafting
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Shu Xu, Attending Physician, General Hospital of Shenyang Military Region
Other Study IDs: GHShenyang_001
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Atherosclerotic Heart Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- atrial fibrillation group: In the case-control trial, patients with atrial fibrillation 7 days after surgery will be assigned to an atrial fibrillation group.
  Interventions: Other: atrial fibrillation
- non-atrial fibrillation group: Patients without atrial fibrillation 7 days after surgery will be assigned to a non-atrial fibrillation group.
  Interventions: Other: non-atrial fibrillation

INTERVENTIONS:
Other: atrial fibrillation — In the case-control trial, patients with atrial fibrillation 7 days after surgery will be assigned to an atrial fibrillation group.
  Groups: atrial fibrillation group
Other: non-atrial fibrillation — In the case-control trial, patients without atrial fibrillation 7 days after surgery will be assigned to a non-atrial fibrillation group.
  Groups: non-atrial fibrillation group

SUMMARY:
To investigate whether apelin can be used as an indicator to predict postoperative atrial fibrillation in patients with coronary atherosclerotic heart disease, and to provide an objective basis for the clinical selection of a preventive intervention program for atrial fibrillation.

DETAILED DESCRIPTION:
Atherosclerosis is a systematic and progressive pathological process, which commonly occurs in the intima of large and medium-sized arteries. The disease can lead to degenerative, proliferative, non-inflammatory lesions; thickening, hardening, and loss of elasticity of the vascular wall, and vascular stenosis; and reduced arterial blood flow. Eventually, organ damage occurs. Coronary atherosclerotic heart disease is the most common chronic degenerative disease caused by atherosclerosis.

Coronary artery bypass grafting (CABG) can effectively increase myocardial blood supply, prevent myocardial infarction, and improve quality of life, and is associated with low rates of surgical complications and mortality. However, new-onset atrial fibrillation is a common complication after coronary artery bypass grafting, with an incidence rate of 30%. It induces hemodynamic instability, is often accompanied by left-ventricular systolic dysfunction and congestive heart failure, and increases the risk of stroke.

Several studies have shown that the initiation and maintenance of atrial fibrillation is strongly associated with inflammation, which affects the electrical and structural remodeling of the heart. The role of C-reactive protein (CRP), a marker of inflammation, has been widely investigated. C-reactive protein is a non-specific acute-phase protein, and is elevated in many cardiovascular diseases, including coronary atherosclerotic heart disease, heart failure and hypertension. Elevated C-reactive protein levels are not only associated with simple and post-surgical atrial fibrillation, but also with cardioversion and recurrence of atrial fibrillation after ablation. However, there is no elevation of C-reactive protein levels in lone atrial fibrillation, indicating that inflammation is associated with cardiovascular disease, but not with atrial fibrillation per se. One of the aims of the present study is to determine how C-reactive protein levels in patients with new-onset atrial fibrillation change after coronary artery bypass grafting.

Apelin has anti-inflammatory effects in different tissues. Ellinor et al. showed that levels of apelin-12 were remarkably low in patients with atrial fibrillation. Recurrence of atrial fibrillation is high in patients with persistent atrial fibrillation and low apelin-12 levels after electrical cardioversion.

Apelin is an endogenous ligand of the G-protein coupled receptor APJ, and exhibits homology to angiotensin II. The signaling system stimulated by apelin regulates many physiological functions and pathological processes. The main target of apelin is the cardiovascular system; it dilates blood vessels, and has antifibrotic and positive inotropic effects. Falcone et al. showed that the risk of recurrence of atrial fibrillation was 3.1 times greater in patients with low apelin levels than those with high apelin levels. Furthermore, Yang et al. concluded that apelin levels were lower in patients with different types of atrial fibrillation than in controls, indicating that apelin might contribute to the initiation and maintenance of atrial fibrillation.

The investigators carried out a literature search on the Web of Science and ClinicalTrials.gov, using the search terms "apelin", "coronary artery bypass", and "atrial fibrillation". The investigators also searched the Wanfang Database and China National Knowledge Infrastructure, using the terms "apelin", "coronary atherosclerotic heart disease", "surgery", and "atrial fibrillation"; or "apelin", "coronary atherosclerotic heart disease", "coronary artery bypass grafting", and "atrial fibrillation". However, the investigators found no clinical studies of the relationship between apelin and atrial fibrillation after coronary artery bypass grafting. The investigators therefore designed the present study to investigate this relationship.

In the cohort study, patients with coronary atherosclerotic heart disease scheduled to undergo coronary artery bypass grafting will be assigned to high and low apelin groups, according to preoperative apelin levels. The incidence of atrial fibrillation will be compared between the two groups 7 days postoperatively. In addition, a case-control trial in the same patients will compare plasma apelin levels and inflammatory response between those patients with and without atrial fibrillation 7 days postoperatively.

Adverse events Adverse events after coronary artery bypass grafting will be recorded. These might include myocardial infarction, myocardial ischemia, bradycardia, hypotension, and stent thrombosis. The investigators will provide a detailed record of date of onset, treatment-related processing method, and possible relationship with treatment. All adverse reactions should be reported to the researcher in charge and clinical Institutional Review Board within 24 hours.

Data collection, management, analysis and open access Data collection: A table will be formulated for data collection according to the trial design. Data will be added to an electronic database using a double data entry strategy.

Data management: Accuracy of information will be checked when all recruited patients are followed up. The database will be locked by the researcher in charge and will not be altered. All information relating to this trial will be preserved by The General Hospital of Shenyang Military Region, China.

Data analysis: The electronic database will be fully disclosed to a statistician for statistical analysis.

Open access: Published data will be available at www.figshare.com.

Statistical analysis Statistical analysis will be performed by a statistician blinded to group assignment, using SPSS 19.0 software. If measurement data are normally distributed, data will be expressed as mean ± SD, and count data will be expressed as percentages. P < 0.05 will be considered statistically significant.

In the cohort study, the chi-square test will be used to compare the incidence rate of new-onset atrial fibrillation after coronary artery bypass grafting in patients with high and low apelin levels.

In the case-control study, paired t-tests will be used to compare plasma apelin, brain natriuretic peptide, and high-sensitivity C-reactive protein levels in patients with and without atrial fibrillation. Multivariate logistic regression analysis will be applied to determine the relationship between plasma apelin levels, cardiac fibrosis and inflammatory response with atrial fibrillation after coronary artery bypass grafting.

Frequency and measures for monitoring trial implementation Trial progression will be reported to the Ethics Committee of the General Hospital of Shenyang Military Region every month and the trial's status will be updated in the registration database.

Confidentiality Test data, including medical records, will be saved electronically and in hard copy. The electronic data will be preserved in a dedicated password-protected computer and managed by a data manager. The paper data will be preserved in a secure, locked place by the data manager and researcher in charge for future viewing.

ELIGIBILITY:
Inclusion Criteria:

* Meet WHO diagnostic criteria for coronary atherosclerotic heart disease
* Are scheduled to undergo coronary artery bypass grafting
* Have no history of atrial fibrillation
* Have no history of thoracotomy
* Provide written informed consent, having understood the benefits and risks of participation in the trial

Exclusion Criteria:

* Valvular heart disease requiring surgical treatment
* Severe cerebrovascular disease
* Malignant tumor
* Severe autoimmune disease
* Thyroid dysfunction
* Severe infection
* Heart failure or acute myocardial infarction in the past month
* Severe dysfunction of the heart, liver or lung
* Refusal to cooperate with specimen collection and laboratory examination
* Ongoing participation in other clinical trials
* Unable to provide informed consent owing to mental disorders or language barriers

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary atherosclerotic heart disease, without a history of atrial fibrillation, and scheduled to undergo CABG. Their baseline data will be assessed according to inclusion and exclusion criteria. Up to 120 patients with coronary atherosclerotic heart disease scheduled to undergo coronary artery bypass grafting (CABG) will be recruited from the Department of Cardiac Surgery, General Hospital of Shenyang Military Region, China.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of new-onset atrial fibrillation | 7 days after surgery

SECONDARY OUTCOMES:
Plasma apelin levels | 7 days after surgery
  Apelin levels in circulating blood are associated with those in the cardiac atrium. Apelin is a cardiovascular polypeptide. The apelin receptor inhibits the angiotensin receptor, and is a protective factor against cardiovascular disease.
Plasma brain natriuretic peptide level | 7 days after surgery
  Atrial fibrillation can cause a marked increase in serum brain natriuretic peptide. Brain natriuretic peptide participates in the onset of atrial fibrillation and can be used to predict its occurrence.
Plasma high-sensitivity C-reactive protein level | 7 days after surgery
  High-sensitivity C-reactive protein(CRP) is a non-specific acute-phase reactive protein, and its levels are elevated in patients with coronary atherosclerotic heart disease, indicating involvement of the inflammatory response.
Cardiac MRI evaluation | 7 days after surgery
  To evaluate the degree of fibrosis of the left and right atrium and pulmonary veins

CONTACTS AND LOCATIONS:
Overall Officials: Shu Xu, Master, Principal Investigator — The General Hospital of Shenyang Military Command, China

IPD SHARING:
Plan to Share IPD: Undecided